CLINICAL TRIAL: NCT06633315
Title: Application of Ketamine Combined With Dexmedetomidine Sedation in Magnetic Resonance Imaging of Children With Autism and Autism Spectrum Disorder:a-Randomized Controlled Trial
Brief Title: Esketamine Combined With Dexmedetomidine Sedation in Head MRI Examination of Children With Autism Spectrum Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maternal and Child Health Hospital of Hubei Province (Other)
Responsible Party: Principal Investigator, Li Na, Deputy chief physician, Maternal and Child Health Hospital of Hubei Province
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MCHH_05
Record Dates: First submitted 2024-09-26; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder; Dexmedetomidine; Esketamine; Sedation
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Dexmedetomidine; Esketamine

STUDY DESIGN:
Intervention Model Description: The children were randomly divided into three groups using a random number table method:
  The low-dose dexmedetomidine group ( DL group,n = 30) ， Group DL received dexmedetomidine 2.5 μ g/kg nasal drops, The high-dose group of dexmedetomidine (DH group),received dexmedetomidine 3 μ g/kg nasal drops The combination group (DE group, n=30). received dexmedetomidine 2 μ g/kg nasal drops plus esketamine 0.5 mg/kg nasal drops.
  Record the Modified Vigilance/Sedation (MOAA/S) Scale score, Mask Acceptance Scale (MAS) score, one-time medication success rate, and number of salvage medication cases 30 minutes after nasal drip. Record the vital signs of four groups of patients during the examination process, including their basic
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose dexmedetomidine (Experimental): received high dose dexmedetomidine,received dexmedetomidine 3 μ g/kg nasal drops,Record the success rate of the first dose of nasal sedation, the onset time of sedation, the time of sedation recovery, the quality of recovery, and the satisfaction of the examining physician. Record the vital signs of three groups of patients during the examination process, including before sedation (T0), after successful sedation (T1), after the end of the examination (T2), and upon awakening (T3). Compare the incidence of adverse reactions during sedation, including bradycardia, nausea and vomiting, nystagmus, postoperative agitation, and delayed awakening, among the three groups of patients.
  Interventions: Other: high dos dexmedetomidine
- Dexmedetomidine and esketamine (Experimental): received dexmedetomidine plus esketamine ,received dexmedetomidine 2 μ g/kg nasal drops plus esketamine 0.5 mg/kg nasal drops.Record the success rate of the first dose of nasal sedation, the onset time of sedation, the time of sedation recovery, the quality of recovery, and the satisfaction of the examining physician. Record the vital signs of three groups of patients during the examination process, including before sedation (T0), after successful sedation (T1), after the end of the examination (T2), and upon awakening (T3). Compare the incidence of adverse reactions during sedation, including bradycardia, nausea and vomiting, nystagmus, postoperative agitation, and delayed awakening, among the three groups of patients.
  Interventions: Other: dexmedetomidine and esketamine
- Low dos dexmedetomidine (Experimental): received dexmedetomidine 2.5 μ g/kg nasal drops, Record the success rate of the first dose of nasal sedation, the onset time of sedation, the time of sedation recovery, the quality of recovery, and the satisfaction of the examining physician. Record the vital signs of three groups of patients during the examination process, including before sedation (T0), after successful sedation (T1), after the end of the examination (T2), and upon awakening (T3). Compare the incidence of adverse reactions during sedation, including bradycardia, nausea and vomiting, nystagmus, postoperative agitation, and delayed awakening, among the three groups of patients.
  Interventions: Other: low dos dexmedetomidine

INTERVENTIONS:
Other: low dos dexmedetomidine — received dexmedetomidine 2.5 μ g/kg nasal drops
  Arms: Low dos dexmedetomidine
Other: high dos dexmedetomidine — received dexmedetomidine 3 μ g/kg nasal drops
  Arms: High dose dexmedetomidine
Other: dexmedetomidine and esketamine — received dexmedetomidine 2 μ g/kg nasal drops plus ketamine 0.5 mg/kg nasal drops
  Arms: Dexmedetomidine and esketamine

SUMMARY:
Objective: To investigate the use of ketamine combined with dexmedetomidine for sedation in children with autism spectrum disorder, Methods:aged 2-6 years,, ASA grade I or II. The children were randomly divided into three groups using a random number table method: a low-dose dexmedetomidine group (DEXL group,n=100）The high-dose group of dexmedetomidine (DEXH group,n=100) and the group of esketamine combined with dexmedetomidine (DEXE group,n=100). The DEXL group received 2.5 μ g/kg of dexmedetomidine nasal drops, the DEXH group received 3 μ g/kg of dexmedetomidine nasal drops, and the DEXE group received 2 μ g/kg of dexmedetomidine nasal drops plus 0.5 mg/kg of ketamine nasal drops. Record the success rate of the first dose of nasal sedation, the onset time of sedation, the time of sedation recovery, the quality of recovery, and the satisfaction of the examining physician. Record the vital signs of three groups of patients during the examination process, including before sedation (T0), after successful sedation (T1), after the end of the examination (T2), and upon awakening (T3).

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD), also known as Autism Spectrum Disorder (ASD), is a condition in which approximately 60% to 70% of autistic children have intellectual disabilities that significantly affect their ability to take care of themselves and bring immense pressure to society and families. Autistic children often have neurological disorders, and therefore require head magnetic resonance imaging (MRI) examinations. MRI examinations can detect abnormal changes in brain structure and function, providing more objective evidence for early diagnosis and valuable treatment time for autistic patients. However, MRI examinations require children to maintain a calm and quiet state, minimizing physical activity as much as possible. Due to the specific interests and behaviors of autistic children, as well as their refusal to accept environmental changes, completing MRI examinations often requires sedation or anesthesia. The main drugs currently used for sedation in pediatric outpatient examinations include dexmedetomidine, midazolam, ketamine, etc. This study aims to select children with ASD who are scheduled to undergo head MRI in outpatient settings, and explore the safety and efficacy of intranasal administration of ketamine combined with dexmedetomidine for sedation, providing reference methods and evidence for sedation in children with autism spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of autism spectrum disorder Aged 2-6 years, ASA grade I or II

Exclusion Criteria:

Upper respiratory tract infections, Severe respiratory system related diseases Congenital heart disease Liver and kidney dysfunction. Contraindications for ketamine and dexmedetomidine, Expected difficult airways. Anesthetic or sedative drugs used in the last week.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
The first success rate of nasal drip | during the procedure
  After the first dose of nasal drip administration, the examination was successfully completed and effective diagnostic images and reports were obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Linli Yue, MD, Principal Investigator — Maternal and Child Health Hospital of Hubei Province
Locations (1):
- Maternal and Child Health Hospital of Hubei Province,, Wuhan, Hubei, China